CLINICAL TRIAL: NCT01861470
Title: Reducing Painful Eye Examinations in Preterm Infants
Brief Title: REDEXAM - Reducing Painful Eye Examinations in Preterm Infants
Acronym: REDEXAM
Status: Completed | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 6650
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm infants: all <32 weeks

SUMMARY:
More than 8000 babies born >8 weeks early or weighing less than 1500g at birth in the United Kingdom annually are at risk of a serious eye problem - retinopathy of prematurity (ROP). Less than 1 in 10 need treating, but to identify these all of them require eye examinations 1-2 weekly from 5 weeks. These tests are uncomfortable, upsetting for families, and cost considerable time and money.

There is now a new urine test that might help identify babies with the highest risk of developing significant ROP. This cheap test appears to predict which babies need treatment and could avoid invasive eye examination in thousands of babies. The test has so far only been used in 136 babies. It accurately predicted ROP, but 136 babies cannot change practice. We need to test more babies including in the UK. This study is designed to test >300 UK babies to see how accurately urine levels of NTproBNP predict development of ROP needing treatment.

We will also pool our data with other researchers across Europe testing the same test to identify the best 'cut'-off' value for this test. In the future babies with urine levels of this chemical lower than this cut-off level would not need invasive eye examinations.

If this test works as we hope it will many babies will avoid repeated painful eye tests, and their families will be saved the stress of watching this being done, by replacing these with a simple easy cheap pain free urine test. There will be substantial savings in health care costs that could be used to improve other aspects of care. In resource poor settings without an expert ophthalmologist babies could be screened for ROP that currently cannot be screened.

We hope to demonstrate this to be a family-friendly, achievable intervention that positively impacts on the lives of babies and families experiencing neonatal intensive care.

DETAILED DESCRIPTION:
See protocol

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants <1500g or <32 weeks gestation

Exclusion Criteria:

* Separate ocular pathology

Max Age: 56 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants <1500g or <32 weeks gestation
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
the ability of urinary NTproBNP (normalised to creatinine) at 14 days of age and 28 days to predict severity of ROP | day 14 and day 28

SECONDARY OUTCOMES:
Receiver operator characteristics curve, sensitivity, specificity, positive and negative predictive values. | day 14 and day 28

CONTACTS AND LOCATIONS:
Overall Officials: Janet Berrington, MD, Principal Investigator — Newcastle-upon-Tyne Hospitals NHS Trust
Locations (1):
- Janet Berrington, Newcastle Neonatal Service, Newcastle, Tyne and Wear, United Kingdom